CLINICAL TRIAL: NCT05468008
Title: Prospective Evaluation of the Clinical Utility of Endoscopic Submucosal Dissection (ESD) in Western Population
Brief Title: Endoscopic Submucosal Dissection (ESD)
Acronym: ESD
Status: Recruiting | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1798539
Record Dates: First submitted 2022-02-23; First posted 2022-07-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Lesion; Barrett Esophagus; Gastrointestinal Lesions
MeSH Terms: conditions — Barrett Esophagus | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — Endoscopic submucosal dissection (ESD) is an outpatient procedure to remove deep tumors from the gastrointestinal (GI) tract

SUMMARY:
This registry is to evaluate the procedural and clinical outcomes in patients undergoing endoscopic submucosal dissection. All patients will receive standard of medical care and no experimental interventions will be performed.

DETAILED DESCRIPTION:
The technique of Endoscopic Mucosal Resection (EMR) is currently widely used in the US to remove precancerous or cancerous lesions confined to the mucosa of the GI tract. EMR carries lower morbidity and mortality compare to surgery, at the expense of a higher rate of piecemeal removal, incomplete resection and cancer recurrence. Endoscopic Submucosal Dissection (ESD) is a newer technique developed in Japan that involves en-bloc resection of the entire lesion irrespective of size, allowing for a detailed analysis of the resected margins and depth of invasion and producing a lower local recurrence. Due to the lack of dedicated ESD devices the procedure has not been disseminated in Western countries. Recently the Food and Drug Administration (FDA) approved a number of devices for ESD. The vast majority of studies evaluating the clinical outcomes from ESD are originating in Japan where the technique is mostly applied to patients with early gastric cancer (Japan has the highest incidence of gastric cancer in the word). In the US lesions that are currently treated with EMR are mostly located in the esophagus (Barrett esophagus) and colon (large adenomatous polyps and intramucosal cancer). These esophageal and colonic lesions can be treated with ESD with expected higher rate of en-block resection and lower recurrence rate compare to EMR. With the differences in patient population and disease location one can anticipate some differences in outcomes between ESD performed in Asian and US patients. Therefore, the investigator wants to prospectively record the experience with ESD done as part of routine medical care in United States (US) population. This will be a prospective data recording study. All patients will receive standard medical care and no experimental interventions will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled to undergo ESD

Exclusion Criteria:

* Any contraindication to performing endoscopy
* Participation in another research protocol that could interfere or influence the outcomes measures of the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the Center of Interventional Endoscopy for standard of care ESD procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the utility of ESD for treatment of gastrointestinal lesions | 12 months
  The primary endpoint of this study will be the prospective evaluation of the utility of ESD for the endoscopic treatment of GI lesions.

SECONDARY OUTCOMES:
En-Bloc Resection Rate | 6 months
  1)This is the proportion of lesions that are resected en-bloc (in one piece) using ESD
Complete Resection Rate | 6 months
  2) This is the proportion of lesions that are completely resected (clean lateral and deep resection margins) with ESD.
Curative Resection Rate | 6 months
  3) This is the proportion of lesions that are considered to have been cured based on endoscopic and histological criteria
Safety- Adverse Events | 12 months
  4) This will be measured based on the rate of adverse events with the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Yang, MD, Principal Investigator — AdventHealth Orlando
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotzev AI, Yang D, Draganov PV. How to master endoscopic submucosal dissection in the USA. Dig Endosc. 2019 Jan;31(1):94-100. doi: 10.1111/den.13240. Epub 2018 Aug 22. PMID 30022521
- [Background] Yang D, Wagh MS, Draganov PV. The status of training in new technologies in advanced endoscopy: from defining competence to credentialing and privileging. Gastrointest Endosc. 2020 Nov;92(5):1016-1025. doi: 10.1016/j.gie.2020.05.047. Epub 2020 Jun 3. PMID 32504699
- [Background] Tanaka S, Kashida H, Saito Y, Yahagi N, Yamano H, Saito S, Hisabe T, Yao T, Watanabe M, Yoshida M, Kudo SE, Tsuruta O, Sugihara KI, Watanabe T, Saitoh Y, Igarashi M, Toyonaga T, Ajioka Y, Ichinose M, Matsui T, Sugita A, Sugano K, Fujimoto K, Tajiri H. JGES guidelines for colorectal endoscopic submucosal dissection/endoscopic mucosal resection. Dig Endosc. 2015 May;27(4):417-434. doi: 10.1111/den.12456. Epub 2015 Mar 5. PMID 25652022
- [Background] Yang D, Othman M, Draganov PV. Endoscopic Mucosal Resection vs Endoscopic Submucosal Dissection For Barrett's Esophagus and Colorectal Neoplasia. Clin Gastroenterol Hepatol. 2019 May;17(6):1019-1028. doi: 10.1016/j.cgh.2018.09.030. Epub 2018 Sep 26. PMID 30267866
- [Background] Yang D, Draganov PV. Expanding Role of Third Space Endoscopy in the Management of Esophageal Diseases. Curr Treat Options Gastroenterol. 2018 Mar;16(1):41-57. doi: 10.1007/s11938-018-0169-z. PMID 29435819
- [Background] Fuccio L, Hassan C, Ponchon T, Mandolesi D, Farioli A, Cucchetti A, Frazzoni L, Bhandari P, Bellisario C, Bazzoli F, Repici A. Clinical outcomes after endoscopic submucosal dissection for colorectal neoplasia: a systematic review and meta-analysis. Gastrointest Endosc. 2017 Jul;86(1):74-86.e17. doi: 10.1016/j.gie.2017.02.024. Epub 2017 Feb 28. PMID 28254526